CLINICAL TRIAL: NCT05010941
Title: Performance of the Hypotension Prediction Index in Living Donor Liver Transplantation
Brief Title: Hypotension Prediction Index in Living Donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2107-228-1240
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-08

CONDITIONS: Living Donor Liver Transplantation; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypotension prediction index: prediction of hypotension events
  Interventions: Device: Hypotension Prediction Index

INTERVENTIONS:
Device: Hypotension Prediction Index — Hypotension Prediction Index monitored via radial arterial line

SUMMARY:
The Hypotension Prediction Index via the Edwards Hemosphere advanced monitoring system is monitored in living donor liver transplantation recipients. The Hypotension Prediction Index is analyzed to verify the performance in predicting hypotensive events.

DETAILED DESCRIPTION:
Hypotensive events during surgery and anesthesia occur frequently and are associated with complications such as myocardial infarction, acute kidney injury, and increase in mortality. Therefore predicting and preventing hypotension can lead to better outcomes.

The Hypotension Prediction Index is monitored with the Edwards Hemosphere advanced monitoring system in living donor liver transplantation recipients via the radial artery. The monitor is blinded so that the anesthesiologist cannot see the index, and the anesthesiologist manages the blood pressure according to the institution's anesthetic protocol for liver transplantation. After the surgery is done, the Hypotension Prediction Index is analyzed to see how well the index predicted actual hypotension that occured during the liver transplantation surgery. Receiver operating characteristic curves are drawn to show the performance of the Hypotension Prediction Index in liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for living donor liver transplantation aged 20 years and older
* Patients who understand the trial and have given informed consent

Exclusion Criteria:

* Patients with arrhythmia or pacemaker

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing living donor liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Prediction of Hypotension 5 Minutes Before the Event | During the surgery
  Receiver operating characteristic curve for the Hypotension Prediction Index, Comparison of the hypotensive event and the Hypotension Prediction Index 5 minutes before the event

SECONDARY OUTCOMES:
Prediction of Hypotension 10 Minutes Before the Event | During the surgery
  Receiver operating characteristic curve for the Hypotension Prediction Index, Comparison of the hypotensive event and the Hypotension Prediction Index 10 minutes before the event
Prediction of Hypotension 15 Minutes Before the Event | During the surgery
  Receiver operating characteristic curve for the Hypotension Prediction Index, Comparison of the hypotensive event and the Hypotension Prediction Index 15 minutes before the event

CONTACTS AND LOCATIONS:
Overall Officials: Hee Soo Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Background] Monk TG, Bronsert MR, Henderson WG, Mangione MP, Sum-Ping ST, Bentt DR, Nguyen JD, Richman JS, Meguid RA, Hammermeister KE. Association between Intraoperative Hypotension and Hypertension and 30-day Postoperative Mortality in Noncardiac Surgery. Anesthesiology. 2015 Aug;123(2):307-19. doi: 10.1097/ALN.0000000000000756. PMID 26083768
- [Background] Sun LY, Wijeysundera DN, Tait GA, Beattie WS. Association of intraoperative hypotension with acute kidney injury after elective noncardiac surgery. Anesthesiology. 2015 Sep;123(3):515-23. doi: 10.1097/ALN.0000000000000765. PMID 26181335
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Davies SJ, Vistisen ST, Jian Z, Hatib F, Scheeren TWL. Ability of an Arterial Waveform Analysis-Derived Hypotension Prediction Index to Predict Future Hypotensive Events in Surgical Patients. Anesth Analg. 2020 Feb;130(2):352-359. doi: 10.1213/ANE.0000000000004121. PMID 30896602
- [Background] Wijnberge M, Geerts BF, Hol L, Lemmers N, Mulder MP, Berge P, Schenk J, Terwindt LE, Hollmann MW, Vlaar AP, Veelo DP. Effect of a Machine Learning-Derived Early Warning System for Intraoperative Hypotension vs Standard Care on Depth and Duration of Intraoperative Hypotension During Elective Noncardiac Surgery: The HYPE Randomized Clinical Trial. JAMA. 2020 Mar 17;323(11):1052-1060. doi: 10.1001/jama.2020.0592. PMID 32065827
- [Background] Maheshwari K, Shimada T, Yang D, Khanna S, Cywinski JB, Irefin SA, Ayad S, Turan A, Ruetzler K, Qiu Y, Saha P, Mascha EJ, Sessler DI. Hypotension Prediction Index for Prevention of Hypotension during Moderate- to High-risk Noncardiac Surgery. Anesthesiology. 2020 Dec 1;133(6):1214-1222. doi: 10.1097/ALN.0000000000003557. PMID 32960954
- [Background] Sudfeld S, Brechnitz S, Wagner JY, Reese PC, Pinnschmidt HO, Reuter DA, Saugel B. Post-induction hypotension and early intraoperative hypotension associated with general anaesthesia. Br J Anaesth. 2017 Jul 1;119(1):57-64. doi: 10.1093/bja/aex127. PMID 28974066
- [Background] Hatib F, Jian Z, Buddi S, Lee C, Settels J, Sibert K, Rinehart J, Cannesson M. Machine-learning Algorithm to Predict Hypotension Based on High-fidelity Arterial Pressure Waveform Analysis. Anesthesiology. 2018 Oct;129(4):663-674. doi: 10.1097/ALN.0000000000002300. PMID 29894315
- [Background] Moller S, Christensen E, Henriksen JH. Continuous blood pressure monitoring in cirrhosis. Relations to splanchnic and systemic haemodynamics. J Hepatol. 1997 Aug;27(2):284-94. doi: 10.1016/s0168-8278(97)80173-0. PMID 9288602
- [Background] Avolio AP, Van Bortel LM, Boutouyrie P, Cockcroft JR, McEniery CM, Protogerou AD, Roman MJ, Safar ME, Segers P, Smulyan H. Role of pulse pressure amplification in arterial hypertension: experts' opinion and review of the data. Hypertension. 2009 Aug;54(2):375-83. doi: 10.1161/HYPERTENSIONAHA.109.134379. Epub 2009 Jun 29. No abstract available. PMID 19564542
- [Background] Shin B, Maler SA, Reddy K, Fleming NW. Use of the Hypotension Prediction Index During Cardiac Surgery. J Cardiothorac Vasc Anesth. 2021 Jun;35(6):1769-1775. doi: 10.1053/j.jvca.2020.12.025. Epub 2020 Dec 21. PMID 33446404
- [Background] Lee HC, Jung CW. Vital Recorder-a free research tool for automatic recording of high-resolution time-synchronised physiological data from multiple anaesthesia devices. Sci Rep. 2018 Jan 24;8(1):1527. doi: 10.1038/s41598-018-20062-4. PMID 29367620